CLINICAL TRIAL: NCT05909007
Title: Post-operative Thoracic Epidural Analgesia and Incidence of Major Complications: a Large Retrospective Dual Center Experi-ence
Status: Completed | Type: Observational
Sponsor: AHEPA University Hospital (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, DESPOINA SARRIDOU, Assistant Professor of Anaesthesia, AHEPA University Hospital
Other Study IDs: 1111
Record Dates: First submitted 2023-06-06; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Neuropathic Pain; Chronic Pain; Thoracic Cancer
MeSH Terms: conditions — Neuralgia; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: thoracic epidural insertion — thoracic epidural for pain relief after major thoracic surgery and lung transplantation

SUMMARY:
A retrospective observational dual center study investigating side effects and major complications after thoracic epidural insertion according to local safety protocols.

DETAILED DESCRIPTION:
Abstract: (1) Background: Thoracic epidural analgesia is considered the gold standard in post-operative pain management following thoracic surgery. This study was designed to explore the safety of thoracic epidural analgesia and to quantify the incidence of its post-operative side-effects in patients undergoing thoracotomy for major surgery, such as resection of lung malignancies and lung transplantation. (2) Methods: This is a retrospective, dual-center observa-tional study implementing patients that underwent major thoracic surgery including lung trans-plantation and received concurrent placement of thoracic epidural catheters for postoperative an-algesia. An electronic system of referral and documentation of complications was used, and information was retrieved from our electronic critical care charting system. Side effects such as nausea and vomiting , itching, catheter related issues and also major complications such as epidural haematoma, abscess, or permanent nerve damage were investigated.

The study aims to highlight the importance of a solid documentation and recording system alongside with the implementation of safety protocols.

ELIGIBILITY:
Inclusion Criteria: 1. All patients undergoing major thoracic surgery ASA1-3 2. All patients undergoing lung transplantation

Exclusion Criteria: 1. Active bleeding 2. Coagulopathy 3. High inflammatory markers 4. SIRS 5. Lack of patients' consent for throracic epidural insertion

-

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients underwent major thoracic surgery and lung transplantation. ASA status 1-3
Sampling Method: Non-Probability Sample
Enrollment: 1145 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
incidence of major complications | 3 YEARS

CONTACTS AND LOCATIONS:
Locations (1):
- Ahepa University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided